CLINICAL TRIAL: NCT04257162
Title: HER2-PREDICT: Translational Study of Tumor Samples From Patients Treated With Trastuzumab Deruxtecan (T-DXd; DS-8201a)
Acronym: HER2-PREDICT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SOLTI Breast Cancer Research Group (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SOLTI-1804; 2019-002991-15 (EudraCT Number)
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Tumor Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Arm (Other): Patients with metastatic cancer treated with Trastuzumab Deruxtecan (T-DXd; DS-8201a)
  Interventions: Other: Tumor and Blood sample collection

INTERVENTIONS:
Other: Tumor and Blood sample collection — This is a non-interventional protocol and does not provide study drug or specific requirements for how the patients should be treated.
  Nevertheless, patients participating in T-DXd trials included in this study are those who were randomized to receive T-DXd.
  Tumor sample and blood sample will be collected within the framework of HER2-Predict Study

SUMMARY:
HER2-Predict is a multi-center, observational study using biological samples from patients treated with DS-8201a in the metastatic setting. Patients will provide a baseline FFPE tumor sample and additionally, blood sample for ctDNA determination will be collected.

ELIGIBILITY:
A. Inclusion Criteria

1. Women and men ≥18 years old that has been included in a trial using Trastuzumab Deruxtecan (T-DXd; DS-8201a).
2. The participant (or legally acceptable representative if applicable) provides written informed consent for the study. It is possible to include patients that were exitus during or after treatment by filling out the appendix 1 form and filing it into the patient's clinical chart.
3. Patients who are starting, are receiving or have received treatment with Trastuzumab Deruxtecan as a treatment for metastatic/advanced cancer.
4. Submission of a formalin-fixed, paraffin-embedded tumor (FFPE) tissue block from the most recently collected tumor tissue, with an associated pathology report, for central molecular analysis and for other protocol-mandated secondary and exploratory assessments. If a newer specimen is either insufficient or unavailable, the patient may still be eligible if the patient can provide a tissue block (preferred) or is willing to consent to and undergo an additional pretreatment core or excisional biopsy (if it is assessable and the biopsy can be safely obtained). The tumor tissue should be of good quality and quantity based on total and viable tumor content.

   1. Acceptable samples include core needle biopsies of the deep metastatic lesion or excisional, incisional, punch, or forceps biopsies for cutaneous, subcutaneous, or mucosal lesions or biopsies from bone metastases.
   2. Fine needle aspiration, brushing, cell pellet from pleural effusion and lavage samples are not acceptable.
5. Patients included before starting experimental treatment must be able and willing to provide blood sample(s).

   B. Exclusion Criteria
6. Not having participated or not willing to participate in a trial using Trastuzumab Deruxtecan.
7. Inability to comply with study and follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-12-13 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
identify the optimal ERBB2 mRNA cut-point predictive of T-DXd response | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (15):
- Spain (15):
  - ICO Badalona, Badalona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Clínic de Barcelona, Barcelona, Barcelona
  - Hospital Universitario de Jerez, Jerez de la Frontera, Cadiz
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Canary Islands
  - H.Univ. Arnau de Vilanova de Lleida, Lleida, Lleida
  - Hospital La Paz, Madrid, Madrid
  - Hospital Virgen de Macarena, Seville, Sevilla
  - Instituto Valenciano de Oncología (IVO), Valencia, Valencia
  - Hospital Universitari Vall d' Hebron, Barcelona
  - ICO Hospitalet, Barcelona
  - Hospital Universitario 12 de octubre, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Virgen del Rocio, Seville

IPD SHARING:
Plan to Share IPD: No